CLINICAL TRIAL: NCT00001362
Title: Structural and Functional Imaging of Neurologically Impaired Patients and Normal Volunteers With 1.5 and 3.0 Tesla MRI
Brief Title: Magnetic Resonance Imaging for the Study of Patients With Neurological Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930060; 93-N-0060
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-07

CONDITIONS: Amnesia; Dementia; Healthy; Nervous System Disease
Keywords: Magnetic Resonance Imaging; Contrast Enhancement; Neuroanatomic Morphometry; Neurobehavioral Deficits; Neurological Disorders; Blood Flow; Blood Volume; Normal Volunteer
MeSH Terms: conditions — Amnesia; Dementia; Nervous System Diseases

SUMMARY:
This study is divided into two parts. The first part of the study will use MRI technology to view the brain structure of patients with neurological disorders and normal volunteers. This portion of the study will attempt to detect specific areas of damage in the brains of patients with amnesia and dementia. It will also try to correlate the amount of brain damage with performance on tests used to measure memory.

In the second part of the study, researchers plan to use MRI technology to study brain function of patients with neurological disorders and normal volunteers when they perform tasks. MRI signals during task performance will be used to record areas of the brain receiving more blood flow indicating increased activity.

Researchers believe this study will help improve existing methods of evaluating patients with neurological disorders. In addition, this study may contribute information about areas of the brain involved in thought processing and motor and sensory function.

DETAILED DESCRIPTION:
We wish to use MRI technology to study brain structure (Part 1) and function (Part 2) in several neurological disorders and in normal controls. In Part 1 of this protocol, we describe our interest in using detailed MRI brain structure analysis to identify predicted specific neural structure atrophy in patients with selective amnesia and dementia and to attempt to associate the magnitude of atrophy in these neural structures with performance on selected memory tests. In Part 2 of this protocol, we outline our interest in utilizing newly developed MRI techniques to identify selective changes in local brain blood volume, blood flow, and other physiological parameters during functional stimulation. Recent developments permit recording of MRI signals that are indicative of regional cerebral blood volume and blood flow changes. Local changes in these physiological measures appear to topographically overlap with expected areas of functional brain activation. The advantage of this method over Positron Emission Tomography is the exquisite spatial resolution of MRI. This MRI technique is new and has had only limited use so far. The studies in Part 2 of this protocol should help develop the method and begin to answer fundamental biological and functional questions about the representation and activation of cognitive, motor, and sensory functions.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects between the ages of 18 and 80.

EXCLUSION CRITERIA:

Patient must be able to give informed consent.

Patients with ferromagnetic objects in their bodies which might be adversely affected by MRI (surgical clips or metal fragments in or near brain, eye or blood vessels, cardiac or neurological pacemaker, cochlear impairments) will be excluded.

Pregnant or lactating women will be excluded. A pregnancy test will be administered to women of childbearing age.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 830
Dates: Start 1992-12; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rueckert L, Lange N, Partiot A, Appollonio I, Litvan I, Le Bihan D, Grafman J. Visualizing cortical activation during mental calculation with functional MRI. Neuroimage. 1996 Apr;3(2):97-103. doi: 10.1006/nimg.1996.0011. PMID 9345480
- [Background] Rueckert L, Appollonio I, Grafman J, Jezzard P, Johnson R Jr, Le Bihan D, Turner R. Magnetic resonance imaging functional activation of left frontal cortex during covert word production. J Neuroimaging. 1994 Apr;4(2):67-70. doi: 10.1111/jon19944267. PMID 8186531
- [Background] Levin HS, Scheller J, Rickard T, Grafman J, Martinkowski K, Winslow M, Mirvis S. Dyscalculia and dyslexia after right hemisphere injury in infancy. Arch Neurol. 1996 Jan;53(1):88-96. doi: 10.1001/archneur.1996.00550010108024. PMID 8599565